CLINICAL TRIAL: NCT06170658
Title: 1 Week Crossover Dispensing Study: Buttermere Versus MiSight 1 Day Soft Contact Lenses
Brief Title: 1 Week Crossover Dispensing Study Between Two Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-23-58
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Lenses, Then Control Lenses (Experimental): Participants will wear the Test Lenses in both eyes for one week and then cross over to the Control Lenses in both eyes for one week.
  Interventions: Device: Test Lenses (stenfilcon A); Device: Control Lenses (omafilcon A)
- Control Lenses, Then Test Lenses (Experimental): Participants will wear the Control Lenses in both eyes for one week and then cross over to the Test Lenses in both eyes for one week.
  Interventions: Device: Test Lenses (stenfilcon A); Device: Control Lenses (omafilcon A)

INTERVENTIONS:
Device: Test Lenses (stenfilcon A) — Daily disposable, silicone hydrogel investigational lenses for one week
Device: Control Lenses (omafilcon A) — Daily disposable, hydrogel commercially available lenses for one week

SUMMARY:
The objective of this investigation is to compare the visual clinical performance of a silicone hydrogel daily disposable investigational contact lenses to a hydrogel daily disposable commercially available contact lenses.

DETAILED DESCRIPTION:
This is a prospective, bilateral, double masked (participant and investigator), randomized, cross-over dispensing study with 1 week wearing period in each arm by comparing visual acuity and subjective vision quality.

ELIGIBILITY:
Inclusion Criteria:

1. Are 8 to 18 years of age inclusive and have full legal capacity to volunteer;
2. Have read and signed and dated the Parental Permission Form (for those aged 16 and younger); participant has read, signed and dated the study Information Consent Letter (if aged 17 or 18 years) or Assent (aged 16 and younger);
3. Are willing and able to follow instructions and maintain the appointment schedule;
4. Are habitual daily wearers of spherical single vision soft contact lenses to correct for distance vision in each eye;
5. Currently wears spherical soft contact lenses or myopia control soft lenses;
6. Have a pair of wearable back-up spectacles;
7. Are willing and able to wear contact lenses for at least 10 hours a day, 6 days a week while in the study;
8. Are myopic with subjective refraction: -0.75D to -7.00D spherical, with an astigmatism ≤ -0.75D in each eye with maximum spherical equivalent anisometropia of 1.00D
9. Are correctable to a visual acuity of +0.10 logMAR or better (in each eye) with sphero-cylindrical subjective refraction;
10. Have clear corneas with no corneal scars or any active ocular disease;
11. Can be fit with the study contact lenses with a power between -0.75 and -7.00 DS; this translates to best corrected vision sphere refraction that vertexes to a CL power between -0.75 and -7.00 (inclusive) at screening visit.
12. Demonstrate an acceptable fit with the study lenses.
13. Demonstrate that they can safely and independently insert and remove contact lenses at the screening/fitting visit;

Exclusion Criteria:

1. Have taken part in another clinical research study within the last 14 days;
2. Are currently habitual wearers of toric lenses.
3. Have worn any rigid contact lenses or ortho-keratology lenses in the past 30 days
4. Are an extended lens wearer (i.e., sleeping with their lenses)
5. Are on ongoing atropine treatment for myopia control
6. Have a difference of > 1.0 D in best vision sphere subjective refraction between eyes;
7. Have amblyopia and/or strabismus/binocular vision problem
8. Have any known active ocular disease, allergies and/or infection;
9. Have a systemic condition that in the opinion of the investigator may affect a study outcome variable;
10. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
11. Have a known sensitivity to the diagnostic pharmaceuticals to be used in the study;
12. Have undergone refractive error surgery or intraocular surgery;
13. Are a member of CORE directly involved in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
High contrast, binocular, distance visual acuity | 7 days
  Distance visual acuity (LogMAR) will be measured using high and low contrast computer-generated acuity charts.

SECONDARY OUTCOMES:
Subjective Vision Quality | 7 days
  Subjective vision quality on 0-100 scale, integer steps (0 = Very poor; 100 = Excellent vision, totally sharp)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD,FCOptom, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada